CLINICAL TRIAL: NCT03284580
Title: Effectiveness of a Home-based Ergonomic Intervention Program on Overall Quality of Life, Health Satisfaction, and Home Ergonomics in Caregivers of Chronic Post-stroke Patients: a Randomized Controlled Clinical Trial
Brief Title: Effectiveness of a Home-based Ergonomic Intervention Program in Caregivers of Chronic Post-stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, José Manuel Pérez Mármol, Principal Investigator, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rehab in carers of post-stroke
Record Dates: First submitted 2017-09-13; First posted 2017-09-15 (Actual); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Stroke; Quality of Life
MeSH Terms: conditions — Stroke | interventions — Caregivers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ergonomic intervention group (Experimental): Ergonomic intervention program at home for caregivers
  Interventions: Other: Ergonomic intervention
- Postural + kinesiotherapy intervention group (Experimental): A postural + kinesiotherapy intervention program at home for caregivers
  Interventions: Other: Postural plus kinesiotherapy intervention program
- Control or conservative group (Other): A conservative intervention by general information for caregivers
  Interventions: Other: Control or conservative intervention

INTERVENTIONS:
Other: Ergonomic intervention — An ergonomic intervention program focused to caregivers, including recommendation about how they should help themself and the patients activities at home.
  Arms: Ergonomic intervention group
Other: Postural plus kinesiotherapy intervention program — An ergonomic intervention program focused to caregivers, including recommendation about how they should help themself and the patients activities at home.
  Other Names: A postural plus kinesiotherapy intervention program, including excercises for caregivers
  Arms: Postural + kinesiotherapy intervention group
Other: Control or conservative intervention — A control or conservative intervention, including general information about stroke disease for the caregivers of these patients
  Arms: Control or conservative group

SUMMARY:
The objective of the present study is to evaluate the effectiveness of two home-based ergonomic intervention programs compared to a control group on the quality of life of caregivers of post-stroke patients

DETAILED DESCRIPTION:
Stroke is a neurological pathology that can cause functional problems and an impairment to perform activities of daily living at home.

For this reason, these patients need the support of a caregiver. Caregivers of post-stroke patients often have also problems with their quality of life because of the care that they must provide. These problems appear mainly during the support tasks in the activities performed at the patient's home.

The objective of the present study is to evaluate the effectiveness of two home-based ergonomic intervention programs compared to a control group on the quality of life of caregivers of post-stroke patients

ELIGIBILITY:
Inclusion Criteria:

* Being caregivers of post-stroke patients
* Being over 18 years old

Exclusion Criteria:

* Being caregiver of patients with other neurological patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-01-08 (Actual); Primary Completion 2017-08-09 (Actual); Study Completion 2017-08-20 (Actual)

PRIMARY OUTCOMES:
Change from WhoQol-Bref at 8 weeks | Eight weeks
  This test measures quality of life
Change from WhoQol-Bref at 16 weeks | Sixteen weeks
  This test measures quality of life

SECONDARY OUTCOMES:
Change from ergonomic evaluation of the domestic environment at 8 weeks | Eight weeks
  This measurement evaluates if domestic environment is ergonomic
Change from ergonomic evaluation of the domestic environment at 16 weeks | Sixteen weeks
  This measurement evaluates if domestic environment is ergonomic

CONTACTS AND LOCATIONS:
Locations (1):
- José Manuel Pérez Mármol, Córdoba, Spain

REFERENCES:
- [Derived] de Araujo Freitas Moreira KL, Abalos-Medina GM, Villaverde-Gutierrez C, Gomes de Lucena NM, Belmont Correia de Oliveira A, Perez-Marmol JM. Effectiveness of two home ergonomic programs in reducing pain and enhancing quality of life in informal caregivers of post-stroke patients: A pilot randomized controlled clinical trial. Disabil Health J. 2018 Jul;11(3):471-477. doi: 10.1016/j.dhjo.2018.01.003. Epub 2018 Feb 13. PMID 29452985